CLINICAL TRIAL: NCT05644132
Title: Thumb Hemi-Arthroplasty With Natural Kinematics (THANKS) Trial
Acronym: THANKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loci Orthopaedics (Industry)
Collaborators: North American Science Associates Ltd. (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: lnDx01
Record Dates: First submitted 2022-11-18; First posted 2022-12-09 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Osteoarthritis Thumb Base Joint
Keywords: Thumb carpometacarpal joint (CMCJ) arthritis; InDx Implant System
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thumb base joint prosthesis (Experimental)
  Interventions: Device: InDx Implant for the carpometacarpal joint

INTERVENTIONS:
Device: InDx Implant for the carpometacarpal joint — Treatment of thumb base joint arthritis with the InDx Implant

SUMMARY:
This clinical trial aims to evaluate the safety and effectiveness of the lnDx Implant in the treatment of thumb base joint arthritis.

This clinical trial hypothesises that implanting the lnDx prosthesis will improve thumb opposition motion, decrease pain and stiffness, and increase grip and pinch strengths of the carpometacarpal joint in patients with thumb base joint arthritis.

Participants will undergo the following measures to assess their clinical performance:

* Hand X-Ray
* Range of Motion - Kapandji opposition score
* Grip strength, lateral pinch and tip pinch
* Visual Analogue Scale (VAS) for Pain
* Quick Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 18 years of age;
* The patient has a confirmed Grade 1-111 osteoarthritis of the CMG joint on clinical examination and X-ray;
* The patient agrees to abstain from enrolment in any other clinical trials that will conflict or interfere with the interpretation of the results of this study, in the opinion of the Investigator, for the duration of the study;
* The patient is able to understand the aims and objectives of the trial and is willing to consent;
* Be willing and able to return for all study-related follow-up procedures;
* If female, is either using contraception or is postmenopausal, or male partner is using contraception; and
* Have been informed of the nature of the study, agreeing to its requirements, and have signed the informed consent approved by the institutional review board/ethics committee.

Exclusion Criteria:

* The patient is <18 years of age;
* The patient is suffering from Rheumatoid Arthritis;
* The patient is suffering from Grade IV osteoarthritis of the CMG joint;
* The patient is suffering post-traumatic arthritis of the CMG joint;
* The patient is a pregnant/lactating female (tested as per institutional requirements);
* Active or latent infection, or sepsis;
* Insufficient quantity or quality of bone and/or soft tissue;
* Metal or polymer material sensitivity;
* Patients who are unwilling or incapable of following postoperative care instructions or protocol requirements;
* Muscular imbalance, peripheral vascular disease that prohibits adequate healing, or a poor soft-tissue envelope in the surgical field, absence of musculoligamentous supporting structures, or peripheral neuropathy;
* Patient with previous thumb surgery;
* In the opinion of the investigator, any medical condition that makes the subject unsuitable for inclusion in the study, including, but not limited to, subjects with a diagnosis of concomitant injury that may interfere with healing; subjects with clinically significant renal, hepatic, cardiac, endocrine, hematologic, autoimmune, or any systemic disease or systemic infection that may make interpretation of the results difficult; subjects who have undergone systemic administration within 30 days prior to implantation of any type of corticosteroid, antineoplastic, immunostimulating, or immunosuppressive agents;
* Comorbidity that reduces life expectancy to less than 36 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Device Survival | Post-op 1 month
  Device surviving in service where survival is a lack of a device failure.
Device Survival | Post-op 2 month
  Device surviving in service where survival is a lack of a device failure.
Device Survival | Post-op 3 month
  Device surviving in service where survival is a lack of a device failure.
Device Survival | Post-op 6 month
  Device surviving in service where survival is a lack of a device failure.
Device Survival | Post-op 12 month
  Device surviving in service where survival is a lack of a device failure.
DASH Scores (Scale: 0-100) | Post-op 3 months
  Disability of Arm, Shoulder and Hand (DASH) questionnaire to assess upper extremity disability and symptoms. Lower scores indicate better outcomes.
DASH Scores (Scale: 0-100) | Post-op 6 months
  Disability of Arm, Shoulder and Hand (DASH) questionnaire to assess upper extremity disability and symptoms. Lower scores indicate better outcomes.
DASH Scores (Scale: 0-100) | Post-op 12 months
  Disability of Arm, Shoulder and Hand (DASH) questionnaire to assess upper extremity disability and symptoms. Lower scores indicate better outcomes.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) Pain Score | Post-op 2 months
  Subjective measure to assess pain. Lower scores indicate better outcomes.
Visual Analogue Scale (VAS) Pain Score | Post-op 3 months
  Subjective measure to assess pain. Lower scores indicate better outcomes.
Visual Analogue Scale (VAS) Pain Score | Post-op 6 months
  Subjective measure to assess pain. Lower scores indicate better outcomes.
Visual Analogue Scale (VAS) Pain Score | Post-op 12 months
  Subjective measure to assess pain. Lower scores indicate better outcomes.
Grip and pinch strength measurements | Post-op 2 months
  Assessment of Grip, Tip Pinch, and Lateral Pinch strength. Higher scores indicate better outcomes.
Grip and pinch strength measurements | Post-op 3 months
  Assessment of Grip, Tip Pinch, and Lateral Pinch strength. Higher scores indicate better outcomes.
Grip and pinch strength measurements | Post-op 6 months
  Assessment of Grip, Tip Pinch, and Lateral Pinch strength. Higher scores indicate better outcomes.
Grip and pinch strength measurements | Post-op 12 months
  Assessment of Grip, Tip Pinch, and Lateral Pinch strength. Higher scores indicate better outcomes.
Kapandji Score | Post-op 2 months
  Assessment of Range of Motion. Higher scores indicate better outcomes.
Kapandji Score | Post-op 3 months
  Assessment of Range of Motion. Higher scores indicate better outcomes.
Kapandji Score | Post-op 6 months
  Assessment of Range of Motion. Higher scores indicate better outcomes.
Kapandji Score | Post-op 12 months
  Assessment of Range of Motion. Higher scores indicate better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Groeninge, Kortrijk, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cootjans K, Vanhaecke J, Dezillie M, Barth J, Pottel H, Stockmans F. Joint Survival Analysis and Clinical Outcome of Total Joint Arthroplasties With the ARPE Implant in the Treatment of Trapeziometacarpal Osteoarthritis With a Minimal Follow-Up of 5 Years. J Hand Surg Am. 2017 Aug;42(8):630-638. doi: 10.1016/j.jhsa.2017.05.007. Epub 2017 Jun 28. PMID 28666676
- [Background] Craik JD, Glasgow S, Andren J, Sims M, Mansouri R, Sharma R, Ellahee N. Early Results of the ARPE Arthroplasty Versus Trapeziectomy for the Treatment of Thumb Carpometacarpal Joint Osteoarthritis. J Hand Surg Asian Pac Vol. 2017 Dec;22(4):472-478. doi: 10.1142/S0218810417500526. PMID 29117844
- [Background] Crisco JJ, Halilaj E, Moore DC, Patel T, Weiss AP, Ladd AL. In Vivo kinematics of the trapeziometacarpal joint during thumb extension-flexion and abduction-adduction. J Hand Surg Am. 2015 Feb;40(2):289-96. doi: 10.1016/j.jhsa.2014.10.062. Epub 2014 Dec 24. PMID 25542440
- [Background] Dahaghin S, Bierma-Zeinstra SM, Ginai AZ, Pols HA, Hazes JM, Koes BW. Prevalence and pattern of radiographic hand osteoarthritis and association with pain and disability (the Rotterdam study). Ann Rheum Dis. 2005 May;64(5):682-7. doi: 10.1136/ard.2004.023564. Epub 2004 Sep 16. PMID 15374852
- [Background] Eecken SV, Vanhove W, Hollevoet N. Trapeziometacarpal joint replacement with the Arpe prosthesis. Acta Orthop Belg. 2012 Dec;78(6):724-9. PMID 23409567
- [Background] Fitzgerald BT, Hofmeister EP. Treatment of advanced carpometacarpal joint disease: trapeziectomy and hematoma arthroplasty. Hand Clin. 2008 Aug;24(3):271-6, vi. doi: 10.1016/j.hcl.2008.03.003. PMID 18675718
- [Background] Borgers A, Verstreken A, Vanhees M, Verstreken F. Primary endoprosthetic replacement of the arthritic CMC-1 joint. Oper Orthop Traumatol. 2021 Jun;33(3):228-244. doi: 10.1007/s00064-021-00713-y. Epub 2021 May 18. PMID 34003322
- [Background] Duerinckx J, Verstreken F. Total joint replacement for osteoarthritis of the carpometacarpal joint of the thumb: why and how? EFORT Open Rev. 2022 May 31;7(6):349-355. doi: 10.1530/EOR-22-0027. PMID 35638603
- [Background] Farkash U, Sakhnini M, Dreyfuss D, Tordjman D, Rotem G, Luria S. Failure Rate and Early Complications of Thumb Carpometacarpal Joint Replacement-A Multicenter Retrospective Study of Two Modern Implant Designs. J Clin Med. 2023 Dec 25;13(1):121. doi: 10.3390/jcm13010121. PMID 38202128
- [Background] Froschauer SM, Holzbauer M, Mihalic JA, Kwasny O. TOUCH(R) Prosthesis for Thumb Carpometacarpal Joint Osteoarthritis: A Prospective Case Series. J Clin Med. 2021 Sep 10;10(18):4090. doi: 10.3390/jcm10184090. PMID 34575201
- [Background] Ghavami A, Oishi SN. Thumb trapeziometacarpal arthritis: treatment with ligament reconstruction tendon interposition arthroplasty. Plast Reconstr Surg. 2006 May;117(6):116e-128e. doi: 10.1097/01.prs.0000214652.31293.23. PMID 16651933
- [Background] Hansen TB, Snerum L. Elektra trapeziometacarpal prosthesis for treatment of osteoarthrosis of the basal joint of the thumb. Scand J Plast Reconstr Surg Hand Surg. 2008;42(6):316-9. doi: 10.1080/02844310802393974. PMID 18991176
- [Background] Haugen IK, Englund M, Aliabadi P, Niu J, Clancy M, Kvien TK, Felson DT. Prevalence, incidence and progression of hand osteoarthritis in the general population: the Framingham Osteoarthritis Study. Ann Rheum Dis. 2011 Sep;70(9):1581-6. doi: 10.1136/ard.2011.150078. Epub 2011 May 27. PMID 21622766
- [Background] Hernandez-Cortes P, Pajares-Lopez M, Robles-Molina MJ, Gomez-Sanchez R, Toledo-Romero MA, De Torres-Urrea J. Two-year outcomes of Elektra prosthesis for trapeziometacarpal osteoarthritis: a longitudinal cohort study. J Hand Surg Eur Vol. 2012 Feb;37(2):130-7. doi: 10.1177/1753193411414505. Epub 2011 Jul 18. PMID 21768213
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Background] Jorheim M, Isaxon I, Flondell M, Kalen P, Atroshi I. Short-term outcomes of trapeziometacarpal artelon implant compared with tendon suspension interposition arthroplasty for osteoarthritis: a matched cohort study. J Hand Surg Am. 2009 Oct;34(8):1381-7. doi: 10.1016/j.jhsa.2009.04.016. Epub 2009 Aug 15. PMID 19683881
- [Background] Kapandji A. [Clinical test of apposition and counter-apposition of the thumb]. Ann Chir Main. 1986;5(1):67-73. doi: 10.1016/s0753-9053(86)80053-9. French. PMID 3963909
- [Background] Klahn A, Nygaard M, Gvozdenovic R, Boeckstyns ME. Elektra prosthesis for trapeziometacarpal osteoarthritis: a follow-up of 39 consecutive cases. J Hand Surg Eur Vol. 2012 Sep;37(7):605-9. doi: 10.1177/1753193412443501. Epub 2012 Apr 4. PMID 22491000
- [Background] Raj S, Clay R, Ramji S, Shaunak R, Dadrewalla A, Sinha V, Shaunak S. Trapeziectomy versus joint replacement for first carpometacarpal (CMC 1) joint osteoarthritis: a systematic review and meta-analysis. Eur J Orthop Surg Traumatol. 2022 Aug;32(6):1001-1021. doi: 10.1007/s00590-021-03070-5. Epub 2021 Jul 9. PMID 34244850
- [Background] SooHoo NF, McDonald AP, Seiler JG 3rd, McGillivary GR. Evaluation of the construct validity of the DASH questionnaire by correlation to the SF-36. J Hand Surg Am. 2002 May;27(3):537-41. doi: 10.1053/jhsu.2002.32964. PMID 12015732
- [Background] Taleb C, Berner S, Mantovani Ruggiero G. First metacarpal resurfacing with polyvinyl alcohol implant in osteoarthritis: preliminary study. Chir Main. 2014 Jun;33(3):189-95. doi: 10.1016/j.main.2014.03.001. Epub 2014 Mar 20. PMID 24880607
- [Background] van Rijn J, Gosens T. A cemented surface replacement prosthesis in the basal thumb joint. J Hand Surg Am. 2010 Apr;35(4):572-9. doi: 10.1016/j.jhsa.2009.12.026. Epub 2010 Feb 24. PMID 20185250
- [Background] Berkhout MJ, Yin Q, Ritt MJPF. Current Trends in Operative Treatment of Scaphotrapeziotrapezoid Osteoarthritis: A Survey among European Hand Surgeons. J Wrist Surg. 2020 Apr;9(2):94-99. doi: 10.1055/s-0039-3402796. Epub 2020 Feb 12. PMID 32257609
- [Background] Zhang Y, Xu L, Nevitt MC, Niu J, Goggins JP, Aliabadi P, Yu W, Lui LY, Felson DT. Lower prevalence of hand osteoarthritis among Chinese subjects in Beijing compared with white subjects in the United States: the Beijing Osteoarthritis Study. Arthritis Rheum. 2003 Apr;48(4):1034-40. doi: 10.1002/art.10928. PMID 12687546